CLINICAL TRIAL: NCT03352921
Title: Efficacy Of Clinical Pilates Exercises İn Desk-Based Workers With Sagital Cervical Disorientation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Cemaliye Hürer, PHYSİOTHERAPİST, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMU
Record Dates: First submitted 2017-11-09; First posted 2017-11-24 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Sagital Cervical Disorientation
Keywords: clinical pilates; exercise; Sagital Cervical Disorientation; Disorientation; Forward Head Posture
MeSH Terms: conditions — Motor Activity; Confusion | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical pilates exercises (Experimental): The experimental group will receive clinical pilates exercise training in group form for 3 weeks a week for 8 weeks. The training will be done 40-50 minutes per one day. The exercise session will be started with a 10 minute warming program, 30 minutes with the core stabilization training and the clinical pilates exercises with the postural alignment exercises will be applied and the exercise session will be ended with the 10 minutes cooling period.
  Interventions: Other: clinical pilates exercises
- Home exercises program (Active Comparator): For 8 weeks the member in comparison group will be ask to do the exercise program 3 days a week at home. This group will receive a program of stretching, strengthening, and posture exercises. All the exercises in the program will be illustrated on a descriptive form with images. In terms of the follow-up during 8-week duration, the individuals will be called frequently and in the interview by the end of the study.
  Interventions: Other: home exercises program

INTERVENTIONS:
Other: clinical pilates exercises — servikal, deep flexor muscles, posture exercsises
  Other Names: exercise program
  Arms: clinical pilates exercises
Other: home exercises program — stretching, strengthening, and posture exercises to reduce functional disability, to relieve the pain and to provide postural straightening.
  Other Names: classical exercises
  Arms: Home exercises program

SUMMARY:
The aim of this study is to compare the effects of clinical pilates exercises and home exercise program on postural disorders, pain intensity, normal range of motion, muscle strength, endurance, muscle shortness, joint position sense and functional status in desk workers with sagittal cervical disorientation.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain at least for three months,
* Anterior head translation of sagittal segmental alignment disorders,
* Craniovertebral angle as <50 degree,
* Desk-work minimum for 3 years,
* Working with the computer daily at least for 5 hours,
* Less severe physical activity level according to the International Physical Activity Questionnaire.

Exclusion Criteria:

* Taken any physiotherapy program for the last 6 months due to neck or back pain complain,
* Pain severe 3 cm or less according to the Visual Analog Scale (VAS),
* Structural scoliosis,
* Broken neck history
* Rheumatic disorder that affects the neck,
* Acute torticollis,
* Vertebral column surgical history,
* Spinal cord compression due to tumor or other reasons,
* Neurological deficit,
* Temporomandibular joint problem,
* Taking any kind of pain killers except for basic analgesics.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Postural Disorders | eigth weeks
  The evaluation of cervical and upper thoracic posture will be done through the lateral photography. A camera placed on the tripod will be placed 1,5 m away from the patient while standing in a standing position, and the lens of the camera corresponds to the shoulder of the person. Before the patients will be asked to be on their neutral position, they will be asked to move their heads forth and back for the three times and leave their two arms loose next to the body. Angular calculations will be done by attaching reflective markers to their anatomical points of T4 spinosus process, C7 spinosus process, tragus and eye canthus before the photography. Computer program (Markus Bader-MB Software Solutions, triangular screen ruler) will be used for the angular calculations (craniovertebral angle, head tilt angle, cervico-thoracic angle).

SECONDARY OUTCOMES:
Cervical Joint Position Sense | 8 weeks
  In order to determine cervical joint position sense, the individual's head will be brought to the target position by the investigator and held for 2 seconds at this position. The individual will be ask to save this position into their minds as it will be remembered later on. Again initial position(0°) will be turned here 10 seconds waiting will be and then in the same position (target position) he or she will be asked to move forward slowly and wait for 2 seconds in the same location. The angular difference between result value and target value will be recorded by reading from the baseline inclinometer. 30 seconds break will be given between measurements (flexion, extension, lateral flexion and rotation). The target position determined for the evaluation of joint position sense of neck flexion and extension is determined as 30°, for left-right lateral flexion is 20° and 30° for left-right rotation. All the tests will be done both eyes open and closed.
Normal Motion of Cervical Joint | 8 weeks
  The cervical normal joint movement will be evaluated by baseline bubble inclinometer. The validity and reliability of the device has been proven and; the active cervical normal joint movements (flexion, extension, left-right lateral flexion, left-right rotation) will be measured.. During sitting, in order to prevent regional movement, the body will be stabilized to the chair with the help of stabilization belt. For each movement, 3 measurements will be done and the best value will be used for the data analysis.
Muscle Strength | 8 weeks
  Hand Held Dynamometer (HHD) will be used for isometric muscle strength measurement of neck muscles. Cervical flexor, extensor, left and right lateral flexors' isometric muscle strength will be evaluated by the dynamometer.Stabilizer Pressure Biofeedback device will be used for muscle strength measurement of M.Longus Kolli, M.Longus Capitis, M. Rectus Capitis Lateralis and M. Rectus Capitis Anterior which are defined as deep cervical flexor muscles.
muscle endurance | 8 weeks
  With the aim of measuring the endurance of neck flexor muscles, the individuals will be asked to lie in the supine position as hands on the abdomen and knees in 90 degrees flexion. 0.5 kg of weight will be placed to the forehead of the patient with the help of a band put above the ears. First the patients will be asked to make cervical retraction and then make a cervical flexion in 10 degrees and the flexion degree will be determined with the help of goniometer.For the evaluation of neck extensor muscle endurance, the individuals will be asked to come up to the chest line and hang their head from the bed while the arms are lying on the side of the body beside the body. There will be weights placed above the ears; 2 kg for women and 4 kg for men.
Neck pain | 8 weeks
  The pain intensity during relaxing and activity of the individuals will be evaluated through VAS. As its validity and reliability has been proven previously the VAS; is the scale which defines the pain intensity on 10 cm line on a horizontal line a "0"= no pain, "10"=severe pain. The individuals will be asked to sign the point on the line which refers to the pain intensity they feel and the distance between "0" point and the signed point will be measured and the numeric value will be recorded as the pain intensity of the individual.
disability scale | 8 weeks
  The first questionnaire - Neck Disability Index- prepared for the neck pain and functional disability can be defined as the adapted version of Oswestry Back Pain Disability Questionnaire applied to the cervical region. The Neck Disability Index evaluates the disability occurred in daily life as a result of neck pain. The Neck Disability Index is composed of 10 items; 4 with subjective symptoms (pain level, head ache, concentration, sleeping) and 6 with daily life activities (personal care, weight lifting, reading, work life, car driving, spare time activities). The pointing is done from 0 to 5.
muscle shortness | 8 weeks
  The sternal and clavicular part of Pectoralis major muscle, M. Pectoralis minor, Adductor and internal rotator (M. Teres major, M. Latissimus dorsi, M. Rhomboideus major and minor) muscle shortness will be evaluated by using a ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurer C, Angin E, Tuzun EH. Effectiveness of clinical Pilates and home exercises in sagittal cervical disorientation: randomized controlled study. J Comp Eff Res. 2021 Apr;10(5):365-380. doi: 10.2217/cer-2020-0186. Epub 2021 Mar 12. PMID 33706543